CLINICAL TRIAL: NCT07111364
Title: Construction of a Deep Learning-Based Precise Diagnostic Framework for Bladder Tumors Using Ultrasound
Brief Title: Construction of a Deep Learning-Based Precise Diagnostic Framework for Bladder Tumors Using Ultrasound: A Multicenter, Ambispective Cohort Study
Acronym: BCA-AI-US
Status: Recruiting | Type: Observational
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BCA-AI-US
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-05

CONDITIONS: Deep Learning; Ultrasound; Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observational diagnostic model development — observational diagnostic model development

SUMMARY:
This study aims to develop an ultrasound image-based deep learning system to enable automatic segmentation, T-staging, and pathological grading prediction of bladder tumors. It seeks to enhance the objectivity, accuracy, and efficiency of bladder cancer diagnosis, reduce reliance on physician experience, and provide support for precision medicine and resource optimization.

ELIGIBILITY:
Inclusion Criteria:① Suspected bladder mass detected by abdominal ultrasound (age ≥18 years);② Patients scheduled for surgical treatment of bladder tumors.

Exclusion Criteria:

* Age >85 years;

  * Patients unable to undergo abdominal/transrectal ultrasound (e.g., uncooperative individuals, technically inadequate images);

    * History of bladder tumor surgery, radiotherapy, chemotherapy, or systemic therapy within 3 months; ④ Patients with indwelling medical devices (e.g., double-J ureteral stents, urinary catheters);

      * Failure to undergo bladder tumor surgery within 2 weeks post-ultrasound; ⑥ Non-urothelial carcinoma or pathologically unconfirmed diagnoses.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study consecutively enrolled patients with suspected bladder tumors prospectively registered at the Department of Urology, Peking University First Hospital and Shanxi Province Cancer Hospital between May 2025 and May 2027.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Overall Diagnostic Accuracy | From may 2025 to may 2027

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided